CLINICAL TRIAL: NCT03370471
Title: Acute Exercise Effects on Word Learning in Aging and Stroke-induced Aphasia
Brief Title: Exercise Effects on Word Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C2238-P
Record Dates: First submitted 2017-10-10; First posted 2017-12-12 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Aging; Aphasia
Keywords: aerobic exercise; learning; language; cognition
MeSH Terms: conditions — Aphasia; Language

STUDY DESIGN:
Intervention Model Description: 2x2 crossover design comparing two learning paradigms (Study Only vs. Retrieval Practice) and two training conditions (Moderate Intensity Exercise vs. Gentle Stretching)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Older Adults (Experimental): Participants complete all four interventions
  Retrieval Practice + Moderate Intensity Exercise: Subjects will engage in 30 minutes of moderate-intensity cycling prior to word learning using Retrieval Practice (active retrieval during learning)
  Retrieval Practice + Gentle Stretching: Subject will engage in 30 minutes of gentle upper- and lower- limb stretching prior to word learning using Retrieval Practice (active retrieval during learning)
  Study Only + Moderate Intensity Exercise: Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)
  Study Only + Gentle Stretching: Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)
  Interventions: Behavioral: Retrieval Practice + Moderate Intensity Exercise; Behavioral: Retrieval Practice + Gentle Stretching; Behavioral: Study Only + Moderate Intensity Exercise; Behavioral: Study Only + Gentle Stretching
- Individuals with Aphasia (Experimental): Participants complete all four interventions
  Retrieval Practice + Moderate Intensity Exercise: Subjects will engage in 30 minutes of moderate-intensity cycling prior to word learning using Retrieval Practice (active retrieval during learning)
  Retrieval Practice + Gentle Stretching: Subject will engage in 30 minutes of gentle upper- and lower- limb stretching prior to word learning using Retrieval Practice (active retrieval during learning)
  Study Only + Moderate Intensity Exercise: Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)
  Study Only + Gentle Stretching: Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)
  Interventions: Behavioral: Retrieval Practice + Moderate Intensity Exercise; Behavioral: Retrieval Practice + Gentle Stretching; Behavioral: Study Only + Moderate Intensity Exercise; Behavioral: Study Only + Gentle Stretching

INTERVENTIONS:
Behavioral: Retrieval Practice + Moderate Intensity Exercise — Subjects will engage in 30 minutes of moderate-intensity cycling prior to word learning using Retrieval Practice (active retrieval during learning)
Behavioral: Retrieval Practice + Gentle Stretching — Subject will engage in 30 minutes of gentle upper- and lower- limb stretching prior to word learning using Retrieval Practice (active retrieval during learning)
Behavioral: Study Only + Moderate Intensity Exercise — Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)
Behavioral: Study Only + Gentle Stretching — Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)

SUMMARY:
The aging Veteran population will substantially increase over the next 10 years, as the 24.9% of Veterans who are currently between 55-64 years of age join the 38.5% who are already over age 65. The risk of stroke more than doubles each decade after age 55, which places Veterans at an ever-increasing risk of suffering stroke-related language impairment (i.e., aphasia). Difficulty retrieving words, which negatively impacts psychosocial well-being and quality of life, is the most common complaint in healthy aging and aphasia. Word retrieval interventions to maintain or restore communicative function are needed. Studies have shown that physical exercise can improve word learning in young adults. This study will investigate the effects of exercise on word learning in aging and aphasia. The results will help the us understand how exercise may be used to optimize word retrieval interventions for our aging Veterans.

DETAILED DESCRIPTION:
Difficulty retrieving the right word to communicate a message is the most common complaint in healthy older adults and individuals with stroke-induced language impairment (i.e., aphasia). Novel word learning paradigms have been used to investigate a variety of behavioral and neuromodulatory approaches to improve word retrieval deficits. Previous novel word learning studies have shown that physical exercise can improve long term recall in healthy young adults and that increased levels of dopamine may be responsible for this effect; however, no studies have investigated the effects of exercise on novel word learning in older adults and individuals with aphasia, and very little is known about the mechanisms that support exercise-enhanced word learning in these populations.

The aims of this study are to:

1) to identify the novel word learning paradigm that facilitates immediate and long-term word recall 2a) to investigate how acute, moderate-intensity exercise alters levels of serum brain-derived neurotrophic factor (BDNF) and plasma dopamine 2b) to describe and quantify the association between novel word learning and any observed changes in serum BDNF and plasma dopamine.

This research will provide a platform for future investigations of immediate exercise effects on word learning, which are essential for achieving our long-term goal of developing exercise-based word retrieval interventions for healthy older Veterans and Veterans with aphasia.

A within subjects crossover design will be used to address Aims 1, 2a and 2b. Subjects will complete aerobic exercise or stretching (training) before engaging in Study Only or Retrieval Practice (learning). Subjects will be counterbalanced within and across conditions. Sixteen healthy older adults (65-89 years) and 16 individuals with aphasia (35-89 years), will be recruited. The study will comprise 18 sessions over 12 weeks. In Week 1, subjects will undergo baseline blood draws, a physical assessment, cognitive and language assessments, and a practice word learning task. In Weeks 2-12, subjects will complete the four conditions. Each condition will last two weeks, with a one-week break between conditions. In each condition, training and learning sessions will take place on Monday, Wednesday and Friday. Training: Subjects will engage in 30 minutes of moderate-intensity cycling or gentle upper and lower limb stretching (control) prior to engaging in a novel word learning task. Learning: Familiar objects (e.g., cup) will be paired with nonwords (e.g., flark). In the Study Only paradigm, object/nonword pairs will be presented three times across three days (Monday, Wednesday, Friday). In the Retrieval Practice paradigm, object/nonword pairs will be presented during the first session (Monday). In subsequent sessions (Wednesday, Friday), subjects will be asked to recall the nonword name of presented objects. Corrective feedback will be provided on each trial. Testing: Recognition and recall testing without corrective feedback will be administered immediately after learning (short-term memory), before training in the second and third learning session (overnight consolidation) and one week after learning (long-term memory). Blood Draws: Three blood samples will be taken at baseline (rest, 30 minutes, 60 minutes). In each of the four conditions, blood samples will be taking during the first and third learning session (at rest, after training, after learning, and 15 minutes after learning). Whole blood will be collected in plain tubes and in anticoagulant-treated tubes for subsequent serum BDNF and plasma dopamine analysis by ELISA. Samples will be analyzed in triplicate to increase reliability.

ELIGIBILITY:
Inclusion Criteria:

* monolingual English speakers
* "low physical activity" on the International Physical Activity Questionnaire
* physician's written approval for participation in moderate-intensity exercise

Exclusion Criteria:

* VO2 max >26 (men) and 22 (women)
* inability to cycle for 3 minutes at 50 revolutions/minute with no resistance
* any comorbid condition with exercise contraindications
* use of hormone replacement therapy

  * dopaminergic
  * anti-depressant
  * anti-psychotic
  * or illicit drugs
* consumption of >14 alcoholic drinks/week or > 1pack of cigarettes/day
* uncorrected hearing or vision impairments that interfere with study procedures
* inability to read or repeat nonwords (e.g., flark)
* inability to learn one novel word during a practice learning task
* below cut-off on the Montreal Cognitive Assessment or the Comprehensive Aphasia Test Cognitive Screen
* and/or >10 on the Beck Depression Inventory

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Rodriguez, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Older Adults | Individuals With Aphasia
Started | 23 | 5
Completed | 16 | 3
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Unable to access veins for blood draw | 0 | 1
Not completed — Screen fail | 1 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the study.
Groups:
- Healthy Older Adults; Individuals With Aphasia: Participants complete all four study interventions
  Retrieval Practice + Moderate Intensity Exercise: Subjects will engage in 30 minutes of moderate-intensity cycling prior to word learning using Retrieval Practice (active retrieval during learning)
  Retrieval Practice + Gentle Stretching: Subject will engage in 30 minutes of gentle upper- and lower- limb stretching prior to word learning using Retrieval Practice (active retrieval during learning)
  Study Only + Moderate Intensity Exercise: Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)
  Study Only + Gentle Stretching: Subjects will engage in 30 minutes of gentle stretching prior to word learning using Study Only (no active retrieval during learning)
- Total: Total of all reporting groups
Arm/Group | Healthy Older Adults | Individuals With Aphasia | Total
Number analyzed (Participants) | 16 | 3 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (5.1) | 57.7 (21.1) | 71.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 9 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 11 | 2 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Study-Specific Word Recall Task
Description: Study-specific word recall task comprising trained items. Participant is shown each trained item and types the name.
  Acquisition: immediately after exercise or stretching on Monday, Wednesday and Friday.
  Consolidation: immediately before exercise or stretching on Wednesday and Friday, one week after training (Friday)
Time Frame: Assessment occurs over a two-week period for each of the 4 intervention/arms: Week 1: Monday, Wednesday, Friday, Week 2: Friday
Measure: Mean (Standard Deviation); unit: number of words gained
Arm/Group | Healthy Older Adults | Individuals With Aphasia
Number analyzed (Participants) | 16 | 3
number of words gained
  Acquisition- Retrieval Practice + Moderate Intensity Exercise | 6.4 (3.6) | 1.7 (2.1)
  Consolidation- Retrieval Practice + Moderate Intensity Exercise | 4.6 (4.1) | 1.5 (2.1)
  Acquisition- Retrieval Practice + Gentle Stretching | 4.8 (3.8) | 1.7 (2.5)
  Consolidation- Retrieval Practice + Gentle Stretching | 4.6 (4.5) | 0.7 (2.1)
  Acquisition- Study Only + Moderate Intensity Exercise | 4.8 (3.6) | 1.7 (3.8)
  Consolidation- Study Only + Moderate Intensity Exercise | 3.6 (3.2) | 1.3 (2.3)
  Acquisition- Study Only + Gentle Stretching | 5.4 (2.7) | 2.7 (2.9)
  Consolidation- Study Only + Gentle Stretching | 3.5 (3.6) | 1.3 (2.3)

2. Secondary Outcome: Serum BDNF Concentration Levels (pg/mL)
Description: Blood samples collected to measure serum BDNF concentration levels (pg/mL), as follows:
  1. Before moderate intensity exercise or gentle stretching
  2. Immediately after moderate intensity exercise or gentle stretching
  3. Immediately after word learning
  4. 15 minutes after word learning
Time Frame: Assessment occurs on Monday, Wednesday and Friday of Week 1 for each of the 4 intervention/arms
Measure: Mean (Standard Deviation); unit: serum BDNF concentration levels (pg/mL)
Arm/Group | Healthy Older Adults | Individuals With Aphasia
Number analyzed (Participants) | 13 | 2
serum BDNF concentration levels (pg/mL)
  Moderate Intensity Exercise- Before Exercise | 195.50 (36.00) | 137.83 (51.88)
  Moderate Intensity Exercise- Immediately After Exercise | 218.98 (79.39) | 156.01 (70.25)
  Moderate Intensity Exercise- Immediately After Learning | 209.95 (75.70) | 153.70 (28.94)
  Moderate Intensity Exercise- 15 Minutes After Learning | 204.17 (57.36) | 129.34 (12.90)
  Gentle Stretching- Before Stretching | 199.92 (48.72) | 180.25 (42.48)
  Gentle Stretching- Immediately After Stretching | 217.14 (49.33) | 201.19 (93.51)
  Gentle Stretching- Immediately After Learning | 222.03 (58.78) | 140.85 (23.66)
  Gentle Stretching- 15 Minutes After Learning | 218.00 (60.00) | 117.76 (40.87)

3. Secondary Outcome: Plasma Dopamine
Description: The investigators will collect blood samples to detect changes in plasma dopamine in the training conditions on Monday and Friday sessions, as follows:.
  1. Before exercise or stretching
  2. Immediately after exercise or stretching
  3. Immediately after word learning
  4. 15 minutes after word learning
Time Frame: Assessment occurs on Monday, Wednesday and Friday of Week 1 for each of the 4 intervention/arms
Population: We were not able to obtain reliable measurements of dopamine for analysis.
Arm/Group | Healthy Older Adults | Individuals With Aphasia
Number analyzed (Participants) | 0 | 0

4. Post Hoc Outcome: Word Recognition
Description: Participants complete word recognition task on trained items.
  Acquisition: immediately after exercise or stretching on Monday, Wednesday, and Friday Consolidation: immediately before exercise or stretching on Monday and Wednesday, and one week after learning (Friday)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of words gained
Arm/Group | Healthy Older Adults | Individuals With Aphasia
Number analyzed (Participants) | 16 | 3
number of words gained
  Acquisition- Retrieval Practice + Moderate Intensity Exercise | 3.1 (2.3) | 4.0 (1.7)
  Consolidation- Retrieval Practice + Moderate Intensity Exercise | 3.0 (3.0) | 3.5 (.07)
  Acquisition- Retrieval Practice + Gentle Stretching | 3.1 (2.0) | 3.0 (3.5)
  Consolidation- Retrieval Practice + Gentle Stretching | 2.9 (2.6) | -1.7 (1.5)
  Acquisition- Study Only + Moderate Intensity Exercise | 2.7 (2.2) | 2.3 (1.5)
  Consolidation- Study Only + Moderate Intensity Exercise | 1.8 (2.4) | 0.3 (2.1)
  Acquisition- Study Only + Gentle Stretching | 1.9 (2.2) | 2.7 (3.1)
  Consolidation- Study Only + Gentle Stretching | 3.2 (2.8) | 1.7 (0.5)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Healthy Older Adults | Individuals With Aphasia
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/5
Other Adverse Events (participants affected / at risk) | 1/23 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Older Adults (N=23) | Individuals With Aphasia (N=5)
Dizziness and Syncope (General disorders) | 1 (1) | 0 (0) — Participant experienced an episode of dizziness and syncope following an exercise session.
Skin Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant spilled coffee while waiting to begin the intervention and experienced redness/burns on skin.

LIMITATIONS AND CAVEATS:
Participants: We were not able to recruit the target number of participants with aphasia. Our small numbers in this arm prevented us from conducting reliable statistical analyses of these data.

Technical problems: We were not able to obtain reliable measurements of dopamine. This hindered completion of our secondary analysis related to the association between word learning and changes in dopamine with exercise and stretching.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT03370471/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT03370471/SAP_001.pdf